CLINICAL TRIAL: NCT02350114
Title: An Observational Study of the Functional Capacity of Heart Failure Patients With Reduced Ejection Fraction Admitted With Acute Heart Failure
Brief Title: An Observational Study of the Functional Capacity of Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Colorado Prevention Center (Other); Cardioxyl Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CXL-AHF-FC01; CV013-007 (Other: BMS)
Record Dates: First submitted 2015-01-18; First posted 2015-01-29 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Acute Heart Failure
Keywords: Heart failure; 6 Minute Walk Test
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Functional Capacity (Experimental): 6 Minute Walk Test
  Interventions: Procedure: 6 Minute Walk Test

INTERVENTIONS:
Procedure: 6 Minute Walk Test — Evaluation of walking distance on standardized 6 minute walk test
  Other Names: Walk Test

SUMMARY:
This is an observational study of the functional capacity of patients with Heart failure with Reduced Ejection Fraction (HFrEF) who are admitted to the hospital for routine medical treatment.

DETAILED DESCRIPTION:
This observational study will evaluate the functional capacity (ability to walk and distance walked) of patients with Heart failure with Reduced Ejection Fraction (HFrEF) in approximately 50-70 patients who present with Acute Heart Failure to approximately 5-6 hospital sites in the USA. All enrolled patients will be evaluated for their baseline functional capacity. Patients will receive standard Acute Heart Failure therapy and will be serially assessed for change in their functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Have a left ventricular ejection fraction (LVEF) ≤40%, as assessed by any method, e.g., echocardiography, a multigated acquisition (MUGA) scan or magnetic resonance imaging (MRI);
* Present with signs and symptoms considered to be primarily due to AHF and be admitted to the hospital for AHF;
* Confirmation verbally that the patient was ambulatory, i.e., able to walk >30m, prior to developing symptoms of AHF leading to the current admission;
* Be capable of understanding the nature of the trial; be willing and able to comply with the inpatient and outpatient study protocol requirements for the duration of the study; and be willing to participate, as documented by written informed consent.

Exclusion Criteria:

* Have a systolic blood pressure <90mmHg or >170mmHg at baseline;
* Have an anticipated need for an invasive procedure within 3 days of study enrollment, e.g., due to hemodynamic or cardiac rhythm instability, or acute coronary syndrome, requiring procedures including, but not limited to, cardiac catheterization, placement of a defibrillator/pacemaker, or placement of a pulmonary artery catheter;
* Have a primary HF etiology attributable to either restrictive/obstructive cardiomyopathy, idiopathic hypertrophic cardiomyopathy (as defined by any wall thickness > 1.8cm) that is obstructive, or uncorrected severe valvular disease (except mitral regurgitation);
* Have any other comorbidities that limit ambulation more than the patient's heart failure, e.g., symptomatic peripheral arterial disease, COPD, arthritis or other condition, as confirmed verbally with the patient;
* Have severe renal insufficiency (defined as a GFR <30mL/min/1.73m2 according to the MDRD equation);
* Have an anticipated survival of less than 90 days, for any reason;
* Have received an investigational agent (drug, device or biologic product) within 30 days (or, if longer, 5 half-lives for a drug or biologic agent) prior to study entry, or be planning to receive an investigational agent at any time throughout the full duration of the study until at least Study Day 35;
* Have any other clinically significant laboratory abnormality, medical condition or social circumstance that, in the investigator's opinion, makes it inappropriate for the patient to participate in this clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Functional Capacity (The 6-minute walk test (6MWT)) | Over up to 5 days of from time of hospitalization
  The 6-minute walk test (6MWT) will be primary measure of functional capacity in these patients.

SECONDARY OUTCOMES:
30-day readmission rates for heart failure | 30 days following discharge from Hospital
  Exploration of the the relationship between 30-day readmission rates for heart failure and functional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: ShiYin Foo, M.D., PhD., Study Director — Cardioxyl Pharmaceiticals
Locations (5):
- United States (5):
  - Cardioxyl Study Site, Indianapolis, Indiana
  - Cardioxyl Study Site, Detroit, Michigan
  - Cardioxyl Study Site, Winston-Salem, North Carolina
  - Cardioxyl Study Site, Cincinnati, Ohio
  - Cardioxyl Study Site, Nashville, Tennessee